CLINICAL TRIAL: NCT04789980
Title: A Multi-center, Prospective, Observational Study to Evaluate Palliative Chemotherapy Patterns and Prognosis in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Good Choice of pALliative Chemotherapy to Patient With Pancreatic Cancer ; GemcitAbine Therapy vs FOLFORINOX therapY
Acronym: GALAXY
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-GTB-OS-401
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer; Palliative Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with locally advanced or metastatic pancreatic cancer who plan to receive palliative chemotherapy

SUMMARY:
The study objectives are to find out: 1) palliative chemotherapy patterns and prognosis in patients with locally advanced or metastatic pancreatic cancer in Korea's real clinical settings, and 2) reasons adopted by clinicians in choosing therapeutic drugs.

DETAILED DESCRIPTION:
This study is a domestic, multi-center, prospective, observational study designed for locally advanced or metastatic pancreatic cancer patients who plan to receive palliative chemotherapy. When patients voluntarily express their consent to provide their information to this study by signing a written agreement, their baseline information including demographics, comorbidities, pancreatic cancer-related information, medical treatment history, etc. shall be used for screening. When patients are judged eligible for study participation, they shall receive an appropriate palliative chemotherapy. After first-line chemotherapy (baseline), information review shall be conducted at month 2, 6 and 12 for chemotherapy currently in use (whether or not chemotherapy ended/discontinued and relevant reasons; type, frequency and duration of administered drugs), RECIST, quality of life (month 2 and 6), activity performance assessment, laboratory tests, tumor marker test, adverse drug reactions, etc. However, if first-line chemotherapy moves to second-line chemotherapy due to causes such as progressive disease (PD), information review shall be restricted to the relevant drug name and survival until the end of the study (month 12).

ELIGIBILITY:
Inclusion Criteria:

1. Patients are briefed about the study objectives and methodologies, and express their consent by signing a written agreement for the use of their personal information.
2. Male and female adults who are ≥ 19 years old at the time of enrollment.
3. Locally advanced or metastatic pancreatic cancer patients whose diagnosis was confirmed histologically or cytologically.
4. Patients who plan to receive palliative chemotherapy (e.g., FOLFIRINOX, Gemcitabine-based therapy, etc.)

Exclusion Criteria:

1. Patients who are diagnosed with any other primary cancer that may influence pancreatic cancer treatment or prognosis.
2. Patients who are currently or have a history of receiving palliative chemotherapy.
3. Female patients who are pregnant, have childbearing potential or are breastfeeding.
4. Patients who are currently participating in other clinical trials (clinical trials for drugs or medical devices) or are planning to participate in other clinical trials during the study period. However, patients participating in a non-interventional observational study or registry study can be enrolled.
5. Other patients who are judged by the investigator to be ineligible to participate in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic pancreatic cancer who plan to receive palliative chemotherapy. Total 1,000 subjects
Sampling Method: Non-Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Chemotherapy patterns(Type of the first-line palliative chemotherapy) | Baseline
  Type of the first-line palliative chemotherapy and reasons for therapy selection/discontinuation
Chemotherapy patterns(Type of the second-line palliative chemotherapy) | up to 12 months
  Type of the second-line palliative chemotherapy for each first-line palliative chemotherapy
Progression-free survival (PFS) | From date of the first tumor response until the date of first documented progression, assessed up to 12 months
  Progression-free survival (PFS) by first-line palliative chemotherapy
Overall Survival (OS) | From date of enrollment until the date of death, assessed up to 12 months
  Overall Survival (OS) by first-line palliative chemotherapy

SECONDARY OUTCOMES:
Total administration period | through the first-line chemotheraphy completion, assessed up to 12 months
  Total administration period of the first palliative chemotherapy.
The best response | through the first-line chemotheraphy completion, assessed up to 12 months
  The best response according to RECIST 1.1 criteria, objective response rate (ORR) and disease control rate (DCR)
Quality of Life Assessment | Baseline, Month 2, Month 6
  Quality of life (FACT-Hep) changes in month 2 and 6 after palliative chemotherapy compared to previous therapy
Eastern Cooperative Oncology Group Performance Status (ECOG PS) scores | Baseline, Month 2, Month 6, Month 12
  Changes in ECOG PS scores at month 2, 6 and 12 after palliative chemotherapy compared to previous therapy. The minimum value is 0 and the maximum value is 5, and higher scores mean a worse outcome.

OTHER OUTCOMES:
Adverse drug reactions(ADR) | From the date of the first-line chemotheraphy started until the end of follow-up(12 months)
  Incidence of adverse drug reactions (ADR) associated with first-line palliative chemotherapy
Serious adverse drug reactions(SADR) | From the date of the first-line chemotheraphy started until the end of follow-up(12 months)
  Incidence of serious adverse drug reactions (SADR) associated with first-line palliative chemotherapy
Adverse drug reactions(ADR) caused delay/discontinuation of planned chemotherapy | From the date of the first-line chemotheraphy started until the end of follow-up(12 months)
  Incidence of ADRs that caused delay/discontinuation of planned chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, South Korea